CLINICAL TRIAL: NCT05996445
Title: A Phase 1, First-in-Human, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Activity of XmAb®662 in Monotherapy or in Combination With Pembrolizumab in Advanced Solid Tumors
Brief Title: A Study of XmAb®662 as Monotherapy or in Combination With Pembrolizumab in Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The Sponsor made a business decision to end the study.
Sponsor: Xencor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XmAb662-01
Record Dates: First submitted 2023-06-23; First posted 2023-08-18 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumors
Keywords: IL-12,; interleukin-12; pembrolizumab; Advanced Solid Tumors; Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Sequential Assignments
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation and Expansion XmAb662 administered as monotherapy (Experimental)
  Interventions: Biological: XmAb662
- Dose Escalation and Expansion XmAb662 administered in combination with pembrolizumab (Experimental)
  Interventions: Biological: XmAb662; Biological: Keytruda® (pembrolizumab)

INTERVENTIONS:
Biological: XmAb662 — Intravenous (IV) administration
Biological: Keytruda® (pembrolizumab) — Intravenous (IV) administration
  Arms: Dose Escalation and Expansion XmAb662 administered in combination with pembrolizumab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics of intravenous administration of XmAb662 monotherapy or in combination with pembrolizumab in subjects with advanced solid tumors and to identify the recommended dose regimen that is safe and biologically effective for XmAb662.

DETAILED DESCRIPTION:
This is a first-in-human (FIH), Phase 1, open-label, multicenter dose escalation study with cohort expansion at one or more recommended dose(s) (RDs), designed to evaluate the safety and tolerability of XmAb662 monotherapy or in combination with pembrolizumab in subjects with selected solid tumors that have progressed after standard/approved therapies, or for which there are no effective available therapies. This study will be conducted in 2 parts: dose escalation (Part 1) and dose expansion (Part 2), and subdivided into arms for XmAb662 monotherapy and XmAb662+pembrolizumab combination.

ELIGIBILITY:
Inclusion Criteria:

Advanced, recurrent or metastatic solid malignancy that is not amenable to curative-intent treatment and which has progressed after standard therapy appropriate for the following tumor type: Head and neck squamous cell carcinoma, melanoma, non-small cell lung cancer, small cell lung cancer (SCLC), urothelial carcinoma, colorectal cancer, gastric cancer, esophageal cancer, cervical cancer, hepatocellular carcinoma, Merkel cell carcinoma, renal cell carcinoma, endometrial cancer, cutaneous squamous cell carcinoma, breast cancer, ovarian cancer (epithelial), castration-resistant prostate cancer (adenocarcinoma)

Measurable disease by RECIST 1.1; subjects with prostate cancer who have evaluable disease according to PCWG3 criteria may enroll

Life expectancy of at least 3 months

Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

For dose escalation cohorts, subjects must have adequate archival tumor sample or willing to provide a fresh tumor

Adequate organ function

Exclusion Criteria:

Receiving treatment with the following therapies: Interleukin (IL)-12 either alone or as part of a treatment regimen; checkpoint inhibitors given within 4 weeks of study drug; other anticancer therapies, including chemotherapy or radiation therapy, given within 4 weeks of the start of study drug (palliative radiation given within a 1-week washout is allowed)

History of allergic or anaphylactic/hypersensitivity reaction to immunotherapy

History of a life-threatening (Grade 4) immune-related adverse event (irAE) related to prior immunotherapy or any prior irAE, regardless of grade

History or evidence of any clinically unstable/uncontrolled disorder, condition, or disease (including, but not limited to, cardiopulmonary, renal, metabolic, hematologic, or psychiatric) other than their primary malignancy

Known active central nervous system involvement by malignant disease; subjects with previously treated brain metastases may participate provided they are radiologically and clinically stable

For subjects receiving pembrolizumab, prior Grade 3 or Grade 4 infusion-related reactions to pembrolizumab, or known hypersensitivity to pembrolizumab

Other protocol defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities (DLTs) | First 3 weeks on treatment for each subject]
  Safety and tolerability as assessed by incidence of DLTs and all available data which will be used to determine the recommend dose(s)
Incidence and severity of treatment emergent adverse events (TEAEs) | Up to 2 years
  Safety and tolerability as assessed by incidence of TEAEs, including clinically significant changes in safety laboratory tests and clinical findings

SECONDARY OUTCOMES:
Characterization of pharmacokinetics | 56 Days
  Measurement of Cmax
Characterization of pharmacokinetics | 56 Days
  Measurement of AUC
Objective response rate | Up to 2 years
  Objective response rate by RECIST 1.1, as modified by PCWG3 for participants with prostate cancer
Progression-free survival | Up to 2 years
  Progression-free survival by RECIST 1.1, as modified by PCWG3 for participants with prostate cancer
Duration of response | Up to 2 years
  Duration of response by RECIST 1.1, as modified by PCWG3 for participants with prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Chet Bohac, MD, Study Director — Executive Medical Director, Clinical Development
Locations (3):
- United States (3):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University Of Virginia Comprehensive Cancer Center, Charlottesville, Virginia